CLINICAL TRIAL: NCT02234609
Title: Effectiveness of Modified Class IV Atraumatic Restorative Treatment - Results After 12 Months
Brief Title: Effectiveness of Modified Class IV Atraumatic Restorative Treatment
Acronym: modARTIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, PD Dr. A. Rainer Jordan, Assistant Professor, University of Witten/Herdecke
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: mARTIV; 76/2011 (Other: Witten/Herdecke IRB)
Record Dates: First submitted 2014-08-25; First posted 2014-09-09 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Dental Caries
Keywords: dentistry; dental caries; atraumatic restorative Treatment; effectiveness
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- adults with incisor dental caries lesion (Other): modified ART class IV with glass ionomer cement
  Interventions: Device: modified ART class IV

INTERVENTIONS:
Device: modified ART class IV — Carious tissue was removed with an excavator until a sound probing was obtained. Restorations were performed using a mechanically improved glass-ionomer cement for ART. The modified class IV ART restoration was inserted into the cavity using a spatula. By these restoration technique, the cavity was (i) sealed to stop further caries progression. The cavity was (ii) capped to protect the vital dentin-pulp-complex from external stimuli. The modified class IV ART was aimed at conserving the carious incisor for prospective functional use and for prolonging tooth preservation rather than at anatomical reconstruction of the tooth form for cosmetic reasons.

SUMMARY:
Atraumatic Restorative Treatment (ART) has become an accepted dental restoration treatment in many developing countries. Because, ART is intended to be operated in molars, and about 10% of all carious lesion by an age of 18 years appear in anterior teeth in Gambia, it was the aim of this study to clinically evaluate a modified ART restoration technique for anterior teeth as the traditional treatment approach did not show satisfying clinical results.

DETAILED DESCRIPTION:
Atraumatic Restorative Treatment (ART) has become an evidence-based treatment in class I caries cavities for countries with developing dental infrastructure. Though epidemiological data also demonstrate restorative treatment needs in anterior teeth in several African countries, scientific evidence for ART in this application appeared so far unrewarding. Consequently, many carious teeth remain untreated or are scheduled for extraction. In deciduous teeth, class III and IV ART presented 86% failures due to partial or complete loss already within the first year, and longitudinal data in the permanent dentition are rare. Survival rates of 71% after three years, and of 68% after six years in the same study cohort were reported from Brazil.

Basically, ART appears to be an interesting treatment approach as it combines a manual cavity preparation technique with the use of a glass-ionomer cement as an adhesive and fluoride releasing restoration material. Biomechanical stress, however, is above-average in class IV restorations when intending to reconstruct the incisal edge with glass-ionomer cement resulting in reported high rates of restoration fractures or loss. It was therefore the aim to evaluate the clinical effectiveness of a modified ART class IV restoration technique in a clinical study. These data are to be compared with an historical control (original ART class IV anatomical structure rebuilding restorations). Historical control data will be retrieved from "Jordan RA, Gaengler P, Markovic L, Zimmer S: Performance of Atraumatic Restorative Tratment (ART) depending on operator-experience. J Public Health Dent 2010; 70: 176-80."

ELIGIBILITY:
Inclusion Criteria:

* informed consent

Exclusion Criteria:

* no class IV cavity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number (and percentage) of class IV modified ART restorations with failures after 1 year of performance (failures are defined as loss of restoration and/or fractures): annual failure rate | 1 year
  Sept 2012 - Sept 2013: participants will be followed-up after 1 year

SECONDARY OUTCOMES:
9 scale clinical evaluation scores of class IV modified ART restorations after 1 year of performance (scores are defined by Frencken et al. 1996): ART evaluation criteria | 1 year
  Sept 2012 - Sept 2013: participants will be followed-up after 1 year ART evaluation criteria were published as follows: "Frencken JF, Makoni F, Sithole W: Atraumatic Restorative Treatment and glas-ionomer sealants in a school oral health programme in Zimbabwe: Evaluation after 1 year. Caries Res 1996, 30:428-433". These index does clinically assess the dental restauration in 1 out of 9 categories from "excellent" to "restoration lost".

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zimmer, Professor, Study Chair — Witten/Herdecke University
Locations (1):
- public dental ward at Kindergarten Wattenscheid in Brikama-Kabafita, West Coast Region of The Republic of The Gambia, Banjul, The Gambia